CLINICAL TRIAL: NCT02691624
Title: Study of the Change of Breast Cancer Patients' Upper Limb Lymphatic Drainage Pathway After Operation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BCRLResearch001
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Lymphedema of Upper Arm
Keywords: Lymphedema of Upper Arm; Breast cancer; Breast cancer-related Lymphedema; Lymphoscintigraphy
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sentinel lymph node biopsy: Patients of the group is diagnosed with breast cancer and receive lymphoscintigraphy before operation, and will receive sentinel lymph node biopsy
- axillary lymph node dissection: Patients of the group is diagnosed with breast cancer and receive lymphoscintigraphy before operation, and will receive axillary lymph node dissection

SUMMARY:
Lymphoscintigraphy is a noninvasive，accurate and effective imaging modality. In this study, it is used to investigate the imaging characteristics of patients'upper limb lymphatic drainage before operation, and the influence of operation on it.

DETAILED DESCRIPTION:
The global burden of breast cancer continues to increase largely because of the aging and growth of the world population. More than 1.38 million women worldwide were estimated to be diagnosed with breast cancer in 2008, accounting for 23% of all diagnosed cancers in women. Given that the 5-year survival rate for breast cancer is now 90%, experiencing breast cancer is ultimately about quality of life. Women treated for breast cancer are facing a life-time risk of developing lymphedema, a chronic condition that occurs in up to 40% of this population and negatively affects breast cancer survivors' quality of life. It's becoming more and more important to do more research on the breast cancer-related lymphedema. Axillary reverse mapping (ARM) is a technique used to map arm lymphatic drainage during axillary lymph node dissection (ALND) and/or sentinel lymph node dissection (SLND). It's necessary for the investigators to understand the participants' upper limb lymphatic drainage before operation and what the investigators have done on it during operation. It can be easy to understand the influence of operation on the participants' upper limb lymphatic drainage, the possibility and safety of reserving lymph nodes draining the upper extremity lymph.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients must fulfil all of the following criteria:

1. Diagnosed with breast cancer
2. There is no metastasis except axillary nodes
3. Agree to receive Lymphoscintigraphy of upper extremity

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Pregnancy or lactation
2. Inflammatory breast cancer
3. Disagree to receive Lymphoscintigraphy of upper extremity
4. History of axillary lymph node resection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 breast cancer patients treated in Peking University People's Hospital Breast Center and agree to receive lymphoscintigraphy of upper extremity.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number and relationship with the sentinel lymph node of lymph nodes containing 99mTc-Dextran injected preoperatively to do upper limb lymphoscintigraphy and resected in the process of the sentinel lymph node biopsy | During operation
  Patients enrolled undertake upper limb lymphoscintigraphy before sentinel lymph node biopsy(SLNB).The lymph nodes draining upper extremity lymph will contain 99mTc-Dextran and can be detected by γ detector during operation. The number and relationship with the sentinel lymph node can be measured.
Number of lymph nodes containing 99mTc-Dextran injected preoperatively to do upper limb lymphoscintigraphy and resected in the process of the axillary lymph node dissection | During operation
  Patients enrolled undertake upper limb lymphoscintigraphy before axillary lymph node dissection(ALND).The lymph nodes draining upper extremity lymph can be detected by γ detector in the tissue resected and axilla after operation. The number of them can be measured.

SECONDARY OUTCOMES:
Pathological result of lymph nodes containing 99mTc-Dextran injected preoperatively to do upper limb lymphoscintigraphy and resected in the process of the sentinel lymph node biopsy | in 5 days after operation
  The pathological result of lymph nodes containing 99mTc-Dextran injected preoperatively to do upper limb lymphoscintigraphy and resected in the process of the sentinel lymph node biopsy will be reported in 5 days after operation
Pathological result of lymph nodes containing 99mTc-Dextran injected preoperatively to do upper limb lymphoscintigraphy and resected in the process of the axillary lymph node dissection | in 5 days after operation
  The pathological result of lymph nodes containing 99mTc-Dextran injected preoperatively to do upper limb lymphoscintigraphy and resected in the process of the axillary lymph node dissection will be reported in 5 days after operation

OTHER OUTCOMES:
Patient upper limb circumference | 1 day before operation and 6 months, 1 year, 1.5year, 2 year, 2.5 year, 3 year, 4 year after operation
  The patients' upper limb circumference will be measured on 1 day before operation and 6 months, 1 year, 1.5year, 2 year, 2.5 year, 3 year, 4 year after operation
Patients' bioimpedence value | 2016-2019
  The bioelectrical impedance measurement was performed during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, Principal Investigator — Peking University People's Hospital Breast Center
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fu MR. Breast cancer-related lymphedema: Symptoms, diagnosis, risk reduction, and management. World J Clin Oncol. 2014 Aug 10;5(3):241-7. doi: 10.5306/wjco.v5.i3.241. PMID 25114841
- [Background] Zhu YQ, Xie YH, Liu FH, Guo Q, Shen PP, Tian Y. Systemic analysis on risk factors for breast cancer related lymphedema. Asian Pac J Cancer Prev. 2014;15(16):6535-41. doi: 10.7314/apjcp.2014.15.16.6535. PMID 25169483
- [Background] Suami H, Taylor GI, Pan WR. The lymphatic territories of the upper limb: anatomical study and clinical implications. Plast Reconstr Surg. 2007 May;119(6):1813-1822. doi: 10.1097/01.prs.0000246516.64780.61. PMID 17440362
- [Background] Pavlista D, Eliska O. Analysis of direct oil contrast lymphography of upper limb lymphatics traversing the axilla -- a lesson from the past -- contribution to the concept of axillary reverse mapping. Eur J Surg Oncol. 2012 May;38(5):390-4. doi: 10.1016/j.ejso.2012.01.010. Epub 2012 Feb 14. PMID 22336143
- [Background] Thompson M, Korourian S, Henry-Tillman R, Adkins L, Mumford S, Westbrook KC, Klimberg VS. Axillary reverse mapping (ARM): a new concept to identify and enhance lymphatic preservation. Ann Surg Oncol. 2007 Jun;14(6):1890-5. doi: 10.1245/s10434-007-9412-x. Epub 2007 May 4. PMID 17479341
- [Background] Borri M, Schmidt MA, Gordon KD, Wallace TA, Hughes JC, Scurr ED, Koh DM, Leach MO, Mortimer PS. Quantitative Contrast-Enhanced Magnetic Resonance Lymphangiography of the Upper Limbs in Breast Cancer Related Lymphedema: An Exploratory Study. Lymphat Res Biol. 2015 Jun;13(2):100-6. doi: 10.1089/lrb.2014.0039. Epub 2015 Mar 16. PMID 25774851
- [Background] Liu NF, Lu Q, Liu PA, Yan ZX, Wu XF. [Comparison study of radionuclide lymphoscintigraphy and dynamic magnetic resonance lymphangiography for the diagnosis of extremity lymphedema]. Zhonghua Zheng Xing Wai Ke Za Zhi. 2011 Jul;27(4):241-5. Chinese. PMID 22097305
- [Background] Liu NF, Lu Q, Liu PA, Wu XF, Wang BS. Comparison of radionuclide lymphoscintigraphy and dynamic magnetic resonance lymphangiography for investigating extremity lymphoedema. Br J Surg. 2010 Mar;97(3):359-65. doi: 10.1002/bjs.6893. PMID 20101589
- [Background] Norman SA, Localio AR, Potashnik SL, Simoes Torpey HA, Kallan MJ, Weber AL, Miller LT, Demichele A, Solin LJ. Lymphedema in breast cancer survivors: incidence, degree, time course, treatment, and symptoms. J Clin Oncol. 2009 Jan 20;27(3):390-7. doi: 10.1200/JCO.2008.17.9291. Epub 2008 Dec 8. PMID 19064976
- [Background] International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema: 2013 Consensus Document of the International Society of Lymphology. Lymphology. 2013 Mar;46(1):1-11. PMID 23930436
- [Derived] Liu S, Wang N, Gao P, Liu P, Yang H, Xie F, Wang S, Liu M, Wang S. Using the axillary reverse mapping technique to screen breast cancer patients with a high risk of lymphedema. World J Surg Oncol. 2020 Jun 1;18(1):118. doi: 10.1186/s12957-020-01886-9. PMID 32482174